CLINICAL TRIAL: NCT04893369
Title: Determining the Effectiveness of the Pain and Disability Drivers Management Model on the Management of Low Back Pain - a Pilot Study
Brief Title: Determining the Effectiveness of the Pain and Disability Drivers Management Model on the Management of Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-3524
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain
Keywords: Pain management; Rehabilitation; Low back pain
MeSH Terms: conditions — Low Back Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Two-arm nonrandomized pragmatic cluster clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participating patients will be blinded to their therapist's allocation. Outcomes assessor will be blinded to the participants' allocation since data will be coded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Low Back Pain and Disability Drivers Management model (Experimental): Participating clinicians in the intervention arm will use the PDDM model to guide assessment and treatment of their patients and data will be collected over a 12-weeks period.
  Interventions: Other: The Low Back Pain and Disability Drivers Management model
- Low back pain clinical practice guidelines (Active Comparator): Participating clinicians in the active comparator arm will perform assessment and treatment of their patients based on the recommendations from the most recent and high-quality clinical practice guidelines (CPGs) and data will be collected over a 12-weeks period.
  Interventions: Other: Low back pain clinical practice guidelines

INTERVENTIONS:
Other: The Low Back Pain and Disability Drivers Management model — PTs assigned to the intervention arm will undergo a one-day training specific to the PDDM model. The objectives of the workshop are 1) to acquire knowledge on the functioning of the PDDM model by identifying the different domains of the model, and the specific elements that are deemed "problematic" for a given patient to appropriately establish the clinical profile and 2) to adopt a structured approach to manage and select appropriate interventions to address problematic areas. The model is composed of five domains upon which the clinician can base his assessment and orientate treatment allocation and includes: 1) nociceptive pain drivers, 2) nervous system dysfunction (NSD) drivers, 3) comorbidity drivers, 4) cognitive-emotional drivers and 5) contextual drivers. This profiling will inform and lead the clinician's treatment approach based on the combined contribution of each domain driving the experience of pain and disability.
  Arms: The Low Back Pain and Disability Drivers Management model
Other: Low back pain clinical practice guidelines — For the PTs allocated to the control arm, they will participate in a three-hour training on the most recent CPGs on the management of LBP. The content of the training is based on the results of a thorough review of the literature summarizing the different recommendations from CPGs with a focus on the rehabilitation management of LBP. The objectives of the workshop are 1) to acquire knowledge about the recommendations from the most recent and high-quality CPGs for the management of LBP and 2) to foster their integration into clinical practice. An interactive workshop will be conducted to present the results of the review of the literature with the help of case-studies to facilitate implementation and promote active participation.
  Arms: Low back pain clinical practice guidelines

SUMMARY:
This study aims to assess the feasibility of procedures for conducting a pragmatic cluster nonrandomized controlled trial and to collect data on the effectiveness of a previously validated approach that takes into account all the pain and disability drivers associated with low back pain - the Pain and Disability Drivers Management Model (PDDM).

The overall objective is to provide data to assess the feasibility of implementing a multisite pragmatic cluster nonrandomized clinical trial to determine the effectiveness of the PDDM on short-term patient-related outcomes compared to the most recent clinical practice guidelines to improve the management of patients living with low back pain.

DETAILED DESCRIPTION:
Rationale: Low back pain (LBP) is highly prevalent, recurrent and is the leading cause of disability among all MSK disorders (1). Evidence endorses the use of clinical practice guidelines (CPGs) to help clinicians establish the diagnosis and guide treatments. Yet, they have shown limitations as they mostly focus on addressing biological deficits and poorly integrate psychosocial factors. Thus, we recently developed and validated the Low Back Pain and Disability Drivers Management (PDDM) model that aims to identify the domains influencing pain and disability to create a personalized clinical profile facilitating diagnosis, prognostic and treatment options (2).

Aims and hypotheses: 1) To assess the feasibility of procedures for conducting a pragmatic cluster nonrandomized controlled trial and 2) to explore preliminary evidence of the effectiveness of the PDDM model compared to CPGs on short-term patient-related outcomes. We hypothesize that the feasibility of conducting such trial will be confirmed. Our secondary hypothesis is that the PDDM model will lead to better short-term patients' outcomes compared to CPGs.

Methods:

Design: A pilot cluster nonrandomized controlled trial where allocation occurs at the level of the clinics (CONSORT). Physiotherapy clinics from different demographic and administrative settings will be recruited.

Participants: We aim to recruit a minimum of 12 physiotherapists (PT) per group arm with each PT recruiting a minimum of 5 patients within a 9-month timeframe. To be included, PTs will have to 1) be working with LBP patients, 2) be able to participate in a 1-day training workshop and 3) assess and initiate treatment of their patients guided by the PDDM model (intervention group) or CPGs (comparator). Patients 18 years or older presenting with a primary complaint of LBP without serious underlying pathology will be included.

Intervention: PTs in the intervention group will undergo a 1-day workshop on the PDDM model. In the control group, PTs will be blinded to the PDDM and will receive a 1-day training on CPGs for LBP.

Outcomes: Feasibility outcome measures will include: 1) feasibility of trial design and procedures, 2) recruitment and retention rates, 3) suitability of eligibility criteria and 4) fidelity of intervention. Feasibility success criteria will be determined to guide the decision on conducting a future definitive trial. Effectiveness outcomes will be measured by validated self-reported questionnaires, and more precisely by changes in severity and impact of pain on function, nervous system dysfunctions, cognitive-affective and contextual drivers at baseline, 6- and 12-week follow-ups.

Analysis: Descriptive statistics will be used to summarize feasibility outcomes. Quantitative analysis will be conducted using linear mixed models to explore between- and within-group differences.

Discussion: This project will lead to a better understanding of LBP management as well as the effectiveness of the PDDM model, which has the potential to influence clinical practice by integrating prognostic factors and innovative clinical tools (e.g., patient dashboard to document clinical profile).

ELIGIBILITY:
Clinicians' eligibility criteria:

Inclusion Criteria:

* be working with patients presenting with LBP
* be able to participate in a one-day training workshop
* assess and initiate treatment of their LBP patients based on the PDDM model (intervention) or the most recent CPGs (control)
* be fluent in French

Exclusion Criteria:

* For the control group, clinicians will be excluded if they have already attended a workshop on the PDDM model

Patients' eligibility criteria:

Inclusion Criteria:

* be 18 years or older
* presenting with a primary complaint of LBP
* be able to understand and read French
* have access to an email address
* be willing to provide patient-related outcomes measures

Exclusion Criteria:

* Patients not deemed fit for rehabilitation by their therapist (i.e., red flags)
* Patients already undergoing physiotherapy treatment for their episode of LBP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited for the study | up to nine months.
  Overall recruitment of participants during the nine months recruitment period. Recruitment rate defined as % of eligible clinicians who enrolled in the study for each clinic. Clinician/patient recruitment ratio.
Retention rate of participants | T2 (12 weeks post enrollment for patients and through study completion, up to nine months for clinicians)
  Measured by attrition rate of the participants : % of patients enrolled in the study but who did not complete the study (e.g., questionnaires, dropped out, lost to follow-up)
Suitability of admissibility criteria | T2 (through study completion, up to nine months)
  Determined based on overall recruitment rate and clinicians' answers to two questions at the end of the study (T2): are the criteria sufficient or too restrictive? Is it obvious who meets and who does not meet the eligibility criteria
Clinicians' compliance to study protocol/fidelity of intervention | T2 (through study completion, approximately nine months)
  Assessment of clinician's compliance to the study protocol will include (yes/no): 1) completion of the knowledge and skills assessment following the workshop, and 2) the reporting of five patients' clinical data by the PT according to the PDDM model or CPGs following their initial assessment at baseline (T0).

SECONDARY OUTCOMES:
Change from baseline in severity and impact of pain on function at 12 weeks | Change in BPI scores at 0, 6 and 12 weeks.
  Measured by scores on the Brief Pain Inventory (BPI). Pain intensity (4 items) and pain interference (7 items). Scale 0 to 10. Final score is the average score for each section. Higher scores mean worse outcome).
Change from baseline in nervous system dysfunctions at 12 weeks | Change in PAINdetect scores at 0, 6 and 12 weeks.
  Measured by scores on the PAIN detect questionnaire (12 items, score ranging from 0 to 35)
Change from baseline in nervous system dysfunctions at 12 weeks | Change in CSI-9 scores at 0, 6 and 12 weeks.
  Measured by scores on the short version of the Central Sensitization Index (CSI-9). It contains 9 items, scores ranging from 0 to 36. Higher scores indicate worse outcomes.
Change from baseline in cognitive-affective drivers of pain and disability at 12 weeks | Change in FABQ-physical activity scores at 0, 6 and 12 weeks.
  Measured by scores on the Fear-Avoidance Beliefs Questionnaire - physical activity subscale (FABQ-PA, 4 items, score ranging from 0 to 24)
Change from baseline in cognitive-affective drivers of pain and disability at 12 weeks | Change in CPSS scores at 0, 6 and 12 weeks.
  Measured by scores on the Chronic Pain Self-Efficacy Scale short version (CPSS, 6 items, mean score ranging from 1 to 10). Higher scores indicate better outcomes.
Change from baseline in cognitive-affective drivers of pain and disability at 12 weeks | Change in SBST scores at 0, 6 and 12 weeks.
  Measured by scores on the Start Back Screening Tool (SBST, 9 items, scores ranging from 0 to 9)
Change from baseline in contextual drivers of pain and disability at 12 weeks | Change in FABQ-W scores at 0, 6 and 12 weeks.
  Measured by score on the FABQ-work subscale (FABQ-W, 7 items, score ranging from 0 to 42). Higher score indicates worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Tousignant-Laflamme, PhD, Principal Investigator — Université de Sherbrooke; Michel Tousignant, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longtin C, Lacasse A, Cook CE, Tousignant M, Tousignant-Laflamme Y. Management of low back pain by primary care physiotherapists using the pain and disability drivers management model: An improver analysis. Musculoskeletal Care. 2023 Sep;21(3):916-925. doi: 10.1002/msc.1742. Epub 2023 Feb 10. No abstract available. PMID 36762893
- [Derived] Longtin C, Decary S, Cook CE, Tousignant M, Lacasse A, Tousignant-Laflamme Y. Optimising management of low back pain through the pain and disability drivers management model: Findings from a pilot cluster nonrandomised controlled trial. Musculoskeletal Care. 2023 Sep;21(3):667-682. doi: 10.1002/msc.1738. Epub 2023 Feb 7. PMID 36749025
- See also: Description: Website (online resource) linked to the study that will be available to the participating clinicians in order to facilitate their use of the PDDM model — https://pddmmodel.wordpress.com/